CLINICAL TRIAL: NCT01606995
Title: Xarelto® on Prevention of Stroke and Non-central Nervous System Systemic Embolism in Patients With Non-valvular Atrial Fibrillation
Brief Title: Xarelto for Prevention of Stroke in Patients With Atrial Fibrillation
Acronym: XANTUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 15914; XA1101 (Other: Company internal)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Stroke; Embolism; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism. Decision regarding dose and duration of treatment made at the discretion of the attending investigator

SUMMARY:
This is an international observational study in patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age with a diagnosis of non-valvular atrial fibrillation who start treatment with rivaroxaban to prevent stroke or non-CNS (Central Nervous System) systemic embolism, and who consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of non-valvular atrial fibrillation who start treatment with rivaroxaban to prevent stroke or non-CNS systemic embolism
Sampling Method: Probability Sample
Enrollment: 6784 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2015-03-06 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Adjudicated major bleeding events | after 1 year or until 30 days after end of rivaroxaban therapy
Safety variables will be summarized using descriptive statistics based on adverse events collection | after 1 year or until 30 days after end of rivaroxaban therapy

SECONDARY OUTCOMES:
All cause mortality | after 1 year or until 30 days after end of rivaroxaban therapy
Adjudicated symptomatic thromboembolic events | after 1 year or until 30 days after end of rivaroxaban therapy
Persistence with rivaroxaban treatment: Reasons for any switch from or interruption of rivaroxaban treatment | after 1 year or until 30 days after end of rivaroxaban therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Multiple Locations, Austria
- Multiple Locations, Belgium
- Multiple Locations, Canada
- Multiple Locations, Czechia
- Multiple Locations, Denmark
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Hungary
- Multiple Locations, Ireland
- Multiple Locations, Israel
- Multiple Locations, Moldova
- Multiple Locations, Netherlands
- Multiple Locations, Norway
- Multiple Locations, Poland
- Multiple Locations, Portugal
- Multiple Locations, Russia
- Multiple Locations, Slovakia
- Multiple Locations, Slovenia
- Multiple Locations, Sweden
- Multiple Locations, Ukraine
- Multiple Locations, United Kingdom

REFERENCES:
- [Derived] Kirchhof P, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ. Causes of death in patients with atrial fibrillation anticoagulated with rivaroxaban: a pooled analysis of XANTUS. Europace. 2024 Jul 2;26(7):euae183. doi: 10.1093/europace/euae183. PMID 38941511
- [Derived] Kirchhof P, Haas S, Amarenco P, Hess S, Lambelet M, van Eickels M, Turpie AGG, Camm AJ; XANTUS Investigators*. Impact of Modifiable Bleeding Risk Factors on Major Bleeding in Patients With Atrial Fibrillation Anticoagulated With Rivaroxaban. J Am Heart Assoc. 2020 Mar 3;9(5):e009530. doi: 10.1161/JAHA.118.009530. Epub 2020 Feb 21. PMID 32079476
- [Derived] Amarenco P, Haas S, Hess S, Kirchhof P, Lambelet M, Bach M, Turpie AGG, Camm AJ. Outcomes associated with non-recommended dosing of rivaroxaban: results from the XANTUS study. Eur Heart J Cardiovasc Pharmacother. 2019 Apr 1;5(2):70-79. doi: 10.1093/ehjcvp/pvy041. PMID 30423165
- [Derived] Kirchhof P, Radaideh G, Kim YH, Lanas F, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ; Global XANTUS program Investigators. Global Prospective Safety Analysis of Rivaroxaban. J Am Coll Cardiol. 2018 Jul 10;72(2):141-153. doi: 10.1016/j.jacc.2018.04.058. PMID 29976287
- [Derived] Camm AJ, Turpie AGG, Hess S, Amarenco P, Lambelet M, Haas S, van Eickels M, Kirchhof P; XANTUS Investigators. Outcomes after catheter ablation and cardioversion in patients with non-valvular atrial fibrillation: results from the prospective, observational XANTUS study. Europace. 2018 Jun 1;20(6):e87-e95. doi: 10.1093/europace/eux127. PMID 29016755
- [Derived] Camm AJ, Amarenco P, Haas S, Hess S, Kirchhof P, Kuhls S, van Eickels M, Turpie AG; XANTUS Investigators. XANTUS: a real-world, prospective, observational study of patients treated with rivaroxaban for stroke prevention in atrial fibrillation. Eur Heart J. 2016 Apr 7;37(14):1145-53. doi: 10.1093/eurheartj/ehv466. Epub 2015 Sep 1. PMID 26330425
- [Derived] Camm AJ, Amarenco P, Haas S, Hess S, Kirchhof P, van Eickels M, Turpie AG. XANTUS: rationale and design of a noninterventional study of rivaroxaban for the prevention of stroke in patients with atrial fibrillation. Vasc Health Risk Manag. 2014 Jul 17;10:425-34. doi: 10.2147/VHRM.S63298. eCollection 2014. PMID 25083135
- See also: Click here to find information for studies related to Bayer products. To find this study enter the NCT number or Bayer Study ID in the search field. — http://clinicaltrials.bayer.com/